CLINICAL TRIAL: NCT04644081
Title: Learning Through Play Plus Culturally Adapted Cognitive Behaviour Therapy for Treating Postnatal Depression and Improving Child Wellbeing in Jos Nigeria: A Pilot Randomised Control Trial
Brief Title: LTP+CaCBT for Treating Postnatal Depression and Improving Child Wellbeing in Jos Nigeria
Acronym: LTP+CaCBT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nottingham Trent University (Other)
Collaborators: University of Manchester (Other); Teesside University (Other); Sheffield Hallam University (Other); University of Jos (Unknown)
Responsible Party: Principal Investigator, Dr Dung Jidong, Senior Lecturer/Lecturer, Nottingham Trent University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0000-0001-5034-0335
Record Dates: First submitted 2020-10-29; First posted 2020-11-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Postnatal Depression
MeSH Terms: conditions — Depression, Postpartum | interventions — Behavior Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LTP+CaCBT (Experimental): The LTP+CaCBT intervention will consist of a total of 12 (social distancing) group training sessions (60-90 minutes) and will deliver two sessions on a weekly basis for six weeks.
  Interventions: Behavioral: LTP; Behavioral: CaCBT
- Treatment as Usual (TAU) (Active Comparator): TAU is the routine care currently available for the treatment of postnatal depression at the primary health care sites of intervention (e.g. antidepressants and other forms of counselling services).
  Interventions: Drug: TAU

INTERVENTIONS:
Behavioral: LTP — LTP is a low-literacy, sustainable programme that will provide depressed mothers with valuable skills on parenting, improve mother-child relation and mental health self-care. This is a research-based activity that enhances postpartum mental health while simultaneously promoting attachment security through building parents' ability to monitor and be sensitive to their children's cues, and thereby, actively involves in their children's mental and physical development.
  Other Names: Learning Through Play
  Arms: LTP+CaCBT
Behavioral: CaCBT — CaCBT adopts 'here and now' problem-solving approach, which involves collaborating with families, active listening techniques, changing negative thinking, and depressive symptoms associated with postnatal depression and other forms of parenting distress.
  Other Names: Cultural adapted Cognitive and Behaviour Therapy
  Arms: LTP+CaCBT
Drug: TAU — TAU is the routine care currently available for the treatment of postnatal depression at the primary health care sites of intervention (e.g. antidepressants and other forms of mental health care).
  Other Names: Treatment as Usual
  Arms: Treatment as Usual (TAU)

SUMMARY:
The project aims to test the feasibility, acceptability, cultural appropriateness and effectiveness of LTP+CaCBT for treating postnatal depression and to enhance the mental health and wellbeing of mothers and their children in the low-income areas of Jos Nigeria. This project also aims to provide primary healthcare workers with culturally sensitive requisite skills and support to embed the proposed intervention into routine care practice and increase access to evidence-based intervention.

DETAILED DESCRIPTION:
Participants who scored 10 or above on Patient Health Questionnaire (PHQ-9) and tested positive for postnatal depression on the Edinburgh Postnatal Depression Scale (EPDS) would be recruited randomly assigned into two groups in each of the four primary health care (PHC) facilities designated for the present study. Groups one will receive the LTP+CaCBT treatment - the intervention will consist of a total of 12 (social distancing) group training sessions (60-90 minutes). Groups two will receive routine treatment as usual (TAU) currently available in the PHC facilities (e.g. antidepressants) in the selected communities. Each group will comprise of approximately 10 mother-child pairs.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above
* A mother with a child (0-3 years)
* Able to provide full consent for their participation
* A resident of the trial catchment areas
* Able to complete a baseline assessment
* Score 10 or above on Patient Health Questionnaire (PHQ-9) and tested positive for postnatal depression on the Edinburgh Postnatal Depression Scale (EPDS).

Exclusion Criteria:

* Less than 18 years
* Medical disorder that would prevent participation in a clinical trial such as Tuberculosis or heart failure
* Temporary residents are unlikely to be available for follow up
* Active suicidal ideation or any other severe mental disorder
* Non-residents of Jos and environs
* Unable to consent
* Patients currently undergoing severe mental health treatment
* Unable to speak English language fluently
* Other significant physical or learning disability

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in postnatal depression is being assessed | Change is being assessed from baseline, end of intervention at 6 weeks and at 12 weeks post-intervention
  Primary outcome measure would be assessed using the Edinburgh Postnatal Depression Scale
Change in postnatal anxiety is being assessed | Change is being assessed from baseline, end of intervention at 6 weeks and at 12 weeks post-intervention
  Primary outcome measure would be assessed using the Generalised Anxiety Disorder (GAD7) scale
Change in health is being assessed | Change is being assessed from baseline, end of intervention at 6 weeks and at 12 weeks post-intervention
  Primary outcome measure would be assessed using the Patient Health Questionnaire (PHQ-9)
Change in social support is being assessed | Change is being assessed from baseline, end of intervention at 6 weeks and at 12 weeks post-intervention
  Primary outcome measures would be assessed using the Oslo Social Support Scale
Change in health-related quality of life is being assessed | Change is being assessed from baseline, end of intervention at 6 weeks and at 12 weeks post-intervention
  Outcome measure would be assessed using the Health-related Quality of Life scale (EuroQoL-5 Dimensions)
Change in service satisfaction is being assessed | Change is being assessed at end of intervention at 6 weeks and at 12 weeks post-intervention
  Outcome measure would be assessed using the brief Verona Service Satisfaction Scale
Change in child physio-emotional development is being assessed | Change is being assessed from baseline, end of intervention at 6 weeks and at 12 weeks post-intervention
  Outcome measure would be assessed using the Ages and Stages Social-Emotional Questionnaire
Change in parenting knowledge of child development is being assessed | Change is being assessed from baseline, end of intervention at 6 weeks and at 12 weeks post-intervention
  Outcome measure would be assessed using the Knowledge of Expectation and Child Development Questionnaire

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Jidong DE, Ike TJ, Taru MY, Pwajok JY, Nwoga CN, Jidong JE, Francis C, Mwankon SB, Haruna K, Dagona Z, Husain N. A multi-centred pilot randomised controlled trial of learning through play plus culturally adapted cognitive behaviour therapy for treating postnatal depression in Nigerian women. Front Psychiatry. 2025 May 5;16:1552406. doi: 10.3389/fpsyt.2025.1552406. eCollection 2025. PMID 40391291